CLINICAL TRIAL: NCT05239078
Title: Comparative Evaluation of Pulpal Anaesthetic Efficacy of Different Anaesthetic Solutions for Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis: a Randomized Double-blind Study
Brief Title: Comparative Evaluation of Pulpal Anaesthetic Efficacy of Different Anaesthetic Solutions for Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Vivek Aggarwal (Other)
Collaborators: SGT DENTAL COLLEGE (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Organization: Jamia Millia Islamia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGTTHESIS
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inferior Alveolar nerve block with 2% lidocaine with epinephrine (Active Comparator): An inferior alveolar nerve block was given with 2% lidocaine with epinephrine
  Interventions: Drug: local anaesthetic injection
- Inferior Alveolar nerve block with 4% articaine with epinephrine (Experimental): An inferior alveolar nerve block was given with 4% articaine with epinephrine
  Interventions: Drug: local anaesthetic injection
- Inferior Alveolar nerve block with 3% plain mepivacaine (Experimental): An inferior alveolar nerve block was given with 3% plain mepivacaine
  Interventions: Drug: local anaesthetic injection

INTERVENTIONS:
Drug: local anaesthetic injection — Inferior alveolar nerve block

SUMMARY:
Pulpal and periapical inflammation and infection can cause tissue pH in the affected region to be lowered which results in less penetration of anesthetic solution in the nerve membrane and hence delays the onset of anesthesia. So, the purpose of this study was to compare the pulpal anesthetic efficacy of lidocaine, articaine, mepivacaine for inferior alveolar nerve block (IANB) in patients with irreversible pulpitis (IP). One hundred and twenty adult patients with IP concerning mandibular molars randomly received IANB with either of the three solutions: 2% lidocaine with epinephrine; 4% articaine with epinephrine; 3% plain mepivacaine. Pain during the endodontic treatment was assessed using a visual analog scale (Heft-Parker VAS). Endodontic treatment was initiated. Success was defined as no or mild pain (pain score≤54mm on Hp VAS) during access preparation and root canal instrumentation. The anesthetic success rates were analyzed with the chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* active pain in a mandibular molar
* prolonged response to cold testing with an ice stick and an electric pulp tester
* absence of any periapical radiolucency on radiographs, except for a widened periodontal ligament
* vital coronal pulp on access opening and ability to understand the use of pain scales

Exclusion Criteria:

* known allergy, sensitivity, or contraindications to any opioid or nonopioid analgesic including aspirin or NSAIDs
* history of active peptic ulcer within the preceding 12 months
* history of bleeding problems or anticoagulant use within the last month
* patients who were pregnant or breast-feeding
* a history of known or suspected drug abuse
* patients who had taken NSAIDs within 12 h before administration of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Anesthetic Success | 15 minutes after the inferior alveolar nerve block
  Pain during the endodontic treatment was assessed using a visual analog scale (Heft-Parker VAS). Success was defined as no or mild pain (pain score≤54mm on Hp VAS) during access preparation and root canal instrumentation.

IPD SHARING:
Plan to Share IPD: No